CLINICAL TRIAL: NCT00631553
Title: Assessment of Changes in Renal Cortical and Medullary Blood Flow by Contrast Ultrasound
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Virginia (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Kambiz Kalantarinia MD Assitant Professor of Medicine, University of Virginia Dept of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 12014
Record Dates: First submitted 2008-02-27; First posted 2008-03-07 (Estimated); Last update posted 2008-08-07 (Estimated); Status verified 2008-08

CONDITIONS: Kidney
MeSH Terms: interventions — perflutren

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: perflutren lipid microspheres — 1.3 ml in 30 ml of saline, infused into vein at 2ml / min and titrated for optimal image quality (not to exceed 10 ml/ min at any time).
  Other Names: Definity

SUMMARY:
The purpose of this study is to determine if contrast enhanced ultrasound (CEU) using microbubbles, is useful in assessing changes in kidney blood flow.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults
* Males and females
* Ages 18-65 years old

Exclusion Criteria:

* Pregnancy or lactation
* H/o kidney disease
* H/o congestive heart failure, ischemic heart disease, severe pulmonary disease or allergy to the drug
* H/o any cardiovascular disease
* Abnormal liver function (liver function tests out of specified ranges)
* Screening urinalysis which indicates infection or inflammation
* Taking regular medications (except for over-the-counter vitamins or hormonal contraceptives.)
* Taking supplements, like protein shakes
* Unwilling or unable to eat chicken (used as protein meal)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2006-06; Study Completion 2009-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Kambiz Kalantarinia, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia Health System, Charlottesville, Virginia, United States